CLINICAL TRIAL: NCT04237766
Title: Safety and Effectiveness of a Physiotherapy Intervention Through Movement Visualization in the Approach of Pain in Patients With Hemophilic Arthropathy. Multicenter Randomized Clinical Study.
Brief Title: Movement Visualization in Patients With Hemophilic Arthropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: He-Mirror
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hemophilia
Keywords: Hemophilic arthropathy; Educative intervention; Pain; Quality of life; Anxiety; Stress
MeSH Terms: conditions — Hemophilia A; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): All patients included in the experimental group should be on prophylactic treatment with factor 8 (FVIII) or factor 9 (FIX) concentrates. Likewise, the factor should be administered on the same day that they receive each movement display therapy treatment sessions. Each session will last approximately 40 minutes, with 7 physiotherapy sessions a week taking place over a period of 4 weeks.
  Interventions: Other: Experimental group
- Control group (No Intervention): Subjects included in the control group will not receive physical therapy through mirror therapy and motion display. They will continue with their usual routine of physical activity and exercise, and with the same pharmacological treatment regimen with factor 8 (FVIII) or factor 9 (FIX) concentrates. At the end of the study period the intervention will be applied under the same conditions as the experimental group, analyzing the overall sample at the end of the study.

INTERVENTIONS:
Other: Experimental group — The intervention will consist of the visualization of the movement through the Mirror Therapy application, or through the reproduction of an immersive 360º video emitted on a mobile device and visualized with virtual reality glasses.
  The movements observed with both technologies will be the same. The knee extension and dorsal ankle flexion movements (quadriceps and triceps sural), together with the elbow flexion (elbow flexors) will be the movements to be performed, based on their functional need (ambulation and feeding, respectively).
  Arms: Experimental group

SUMMARY:
Background. The recurrence of hemarthrosis in patients with hemophilia favors the development of an intra-articular, degenerative and progressive lesion (hemophilic arthropathy). Pain is one of the main clinical manifestations of this arthropathy.

Objective. Assess the safety and efficacy of an intervention in pain through visualization of the movement using a mobile application of augmented reality and immersive 360º video, regarding the frequency of bleeding and the improvement of pain perception and quality of life, joint state , strength and functionality in patients with hemophilic arthropathy.

Study design. Randomized, multicenter, simple blind clinical study.

Method. 140 patients with hemophilia A and B will be recruited in this study. Patients will be recruited in 5 regions of Spain. The 8 dependent variables will be: frequency of bleeding (self-registration), pain (measured with the visual analogue scale and pressure algometer, Tampa Scale of Kinesiophobia and Pain Catastrophizing Scale), quality of life (SF-12 scale), anxiety (questionnaire Anxiety State-Trait-STAI), joint state (Hemophilia Joint Health Score scale), muscular strength (dynamometer) and functionality (6-Minutes Walking test, Quick Disabilities of the arm, shoulder and hand). Three evaluations will be carried out: pre-treatment, post-treatment and after a 6-month follow-up period.

Expected results. Observe the effectiveness of movement visualization in the characteristics of pain, and its implication in functionality, joint state, muscular strength and the perception of quality of life in patients with hemophilic arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* Medical diagnosis of hemophilic arthropathy
* Chronic joint pain
* Over 18 years
* On prophylactic treatment or on demand with FVIII / FIX concentrates

Exclusion Criteria:

* Patients with neurological or cognitive disorders that impede the understanding of the questionnaires
* Painless patients
* Amputee, epileptic or seriously impaired vision patients
* Patients receiving physiotherapy treatment at the time of the study
* Patients who have not signed the informed consent document.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline joint bleeding frequency after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  A self-registration of hemorrhages will be used to assess the frequency of bleeding, and with it the safety of the technique. In the self-registration of bleeding, which will be delivered to each patient at the beginning of the study, the patient must fill in the number of hemarthrosis and the main characteristics of these: date, origin (traumatic or spontaneous) and location (knee, ankle or elbow). The self-registration will be delivered to the evaluator in each of the evaluations of the study (post-treatment and follow-up).

SECONDARY OUTCOMES:
Change from baseline joint pain after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The visual analogue scale will be used to assess the perception of joint pain, assessing with a range of 0 to 10 points (from no pain to the maximum pain suffered or imaginable) ankle joint pain.
Change from baseline joint pain perception after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  With a pressure algometer (model Wagner, Wagner Instruments, CT, USA). We will measure pain at pressure, both at the articular level and at a distance (in another part of the body) of patients with hemophilic arthropathy. This device measures in Newton / cm2 the pressure at which the subject perceives pain at the pressure. A pressure will be made on the chosen point, which will increase at an approximate speed of 50 kilopascal / s until the patient warns us that the sensation begins to be painful.
Change from baseline muscle strength after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  With a pressure hand dynamometer the strength of the brachial biceps, quadriceps and sural triceps muscles will be measured. This device measures in Newton the force that the patient performs in the requested muscular action. The higher the value, the greater the muscular strength. We will perform the measurements bilaterally. In measuring the strength of all the muscles evaluated, the average value of the 4 measurements obtained will be used as a measure.
Change from baseline electrical muscle activity after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  Using surface electromyography we will evaluate the electrical activity of the musculature and its activation level. The placement of the electrodes will be marked on the standing subjects, and will be placed following the European recommendations for the use of the surface electromyography. A bipolar surface electromyography system with circular electrodes of 10 mm in diameter, 20 mm apart, placed longitudinally, in the direction of the fibers of the studied muscle, and with a remote reference electrode will be used. A baseline measurement will be performed before the intervention and another during the movement visualization in order to measure the change. The unit of measure is microvolts (µV). The higher the score, the greater the muscular activation.
Change from baseline perception of quality of life after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The perception of quality of life of the patients included in the study will be measured with the Short Form 12 questionnaire (SF-12v2). It consists of 12 items and a range of 0 to 100 points (where a higher score indicates a better perception of quality of life).
Change from baseline anxiety perception after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The anxiety perception of the patients included in the study will be measured with the State-Trait Anxiety Inventory (STAI) questionnaire. The state and anxiety trait of each subject is evaluated with a score of 0 to 30 points for each scale, where a higher score indicates a higher index of anxiety in the trait or state.
Change from baseline fear of movement after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  We will measure the fear of movement of the patients included in the study with the Tampa Scale of kinesiophobia (TSK-11SV) questionnaire. It consists of 11 items. Their values have a range of 1 to 4 points, where the higher the score, the greater the fear of movement.
Change from baseline catastrophism after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  We will measure the catastrophism of the patients included in the study with the Pain catastrophizing scale questionnaire. The scale, composed of 13 items, is valued with a range of 0 to 4 points (lower score indicates lower catastrophism).
Change from baseline anxiety perceived after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The anxiety perceived by the patients included in the study at the time of the intervention will be measured with the Subjective Units of Discomfort Scales questionnaire. This scale, graduated from 0 to 100 where 100 indicates the worst anxiety or discomfort lived or imaginable by the subject, consists of anchored scale a 100mm line will be used where the corresponding value will be marked.
Change from baseline endogenous pain inhibitory system after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The evaluation of the endogenous pain inhibitory system, by facilitating or inhibiting the responses to a conditioned stimulus, will be measured with the Conditioned Pain Modulation Index (CPMI). To perform the evaluation of the diffuse descending inhibitor system, tonic pain will occur by pressing on a non-painful area. First, we will measure the threshold of pain at pressure at the base of the dorsal part of the distal phalanx of the thumb, and then we will cause the conditioned stimulus using the ischemia test on the contralateral upper limb. In this case, for the ischemia test, a sphygmomanometer will be used that will be placed in the arm about 14 cm from the ulnar fossa. The sphygmomanometer will inflate to 240 mmHg and the arm will be placed horizontally.
Change from baseline joint status after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The joint status of patients with hemophilic arthropathy will be measured with the Hemophilia Joint Health Score. This specific scale for use in patients with hemophilia evaluates 8 items: inflammation and duration, pain, atrophy and muscle strength, crepitations, and loss of flexion and extension. It has a score of 0 (no joint damage) to 20 points (maximum joint damage) per joint (elbows, knees and ankles). To the 120 points a gait rating is added (range 0-4 points), the maximum rating of this scale being 124 points.

IPD SHARING:
Plan to Share IPD: No